CLINICAL TRIAL: NCT06287658
Title: The Effect of Kegel Exercise and Ba Duan Jin Applications on Quality of Life and Psychological Well-Being Applied to Premenopausal Women With Urinary Incontinence
Brief Title: The Effect of Kegel Exercise and Ba Duan Jin Applications on Premenopausal Women With Urinary Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Birsen ALTAY, Associate Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-57428665-050.04-240046
Record Dates: First submitted 2024-02-19; First posted 2024-03-01 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Urinary Incontinence; Menopause; Wolman Disease; Quality of Life; Psychological Well-Being
MeSH Terms: conditions — Urinary Incontinence; Wolman Disease; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Kegel exercises and Ba Duan Jin applications will be applied to women in the experimental group online (via Zoom application) in two sessions per week for a total of 8 weeks. Afterwards, women will be asked to perform these practices three days a week for 12 weeks and will be monitored. The research will last a total of 16 weeks.
  Interventions: Behavioral: Training on Kegel exercise and Ba Duan Jin applications online
- Control (Active Comparator): Women in the control group will be given training on Kegel exercises and Ba Duan Jin applications after the research is completed.
  Interventions: Behavioral: training on Kegel exercises and Ba Duan Jin applications after the research is completed

INTERVENTIONS:
Behavioral: Training on Kegel exercise and Ba Duan Jin applications online — Kegel exercises and Ba Duan Jin applications online
  Arms: Experimental
Behavioral: training on Kegel exercises and Ba Duan Jin applications after the research is completed — Women in the control group will be given training on Kegel exercises and Ba Duan Jin applications after the research is completed.
  Arms: Control

SUMMARY:
This study aimed to determine the effects of Kegel exercise and Ba Duan Jin applications applied to premenopausal women with urinary incontinence on quality of life and psychological well-being. Study Group of the Research: Premenopausal women between the ages of 45-55 who come to the family health center with any complaint and have urinary incontinence. The research will be conducted as a randomized pre-test, post-test and control group intervention study design. The research will be conducted with women aged 45-55 with urinary incontinence who came for examination for any reason to a Family Health Center in Sinop between March 2024 and July 2024. According to the power analysis, the number of participants was calculated to be at least 54 when the type 1 error was taken as 0.05, the power was 0.95 and the effect size was medium (0.25) for the two-group design with two repeated measurements. To prevent possible data loss, the sample size was increased by 10% and the total number of participants was determined as 60. A total of 60 women, 30 experimental and 30 control, coming to the Family Health Center will be randomly included in the study. No information, Kegel exercise program and Ba Duan Jin applications will be given to the women in the experimental group, and no intervention will be given to the control group during the research process. Participants will be assigned to 2 groups: experimental and control. Those who come to FHC on odd days of the month will be included in the experimental group, and those who come on even days of the month will be included in the control group. Each group will be determined as 30 people. After the research is completed, the interventions applied to the experimental group will be applied to the women in the control group. Personal Information Form, Psychological Well-Being Scale and Incontinence Quality of Life Scale will be applied to women in the experimental and control groups as pre-test measurements. As a final test, the same measurements will be made to both the control group and the experimental group 16 weeks after the first measurement.

DETAILED DESCRIPTION:
All applications regarding Kegel exercise and Ba Duan Jin applications have been determined. Kegel exercise content; At the beginning of the exercise, one should try to hold urine while emptying the bladder only once or twice in order to define the pelvic floor muscles correctly. If the result is successful, it means that the correct muscles contracted. The second stage, the beginning of the exercise; It can be performed in a supine position (with legs bent at the knee) or in a sitting position. The bladder should be emptied before starting exercise. In the determined position, the pelvic floor muscles should be contracted for 5 seconds, as if stopping urine or gas outflow, and then relaxed for 5 seconds. It should be repeated 4-5 times in a row. The gluteal, abdominal and thigh muscles should not contract. In this way, it is defined that the correct muscles are contracting. In the Ba Duan Jin practice: stretch the hands to the sky, pull the arrow and string the bow (the knees are bent, the sitting posture on the horse is taken, the hand and arm take a stance as if pulling an arrow to the right and left alternately, eyes look at the target in the distance), push the sky and the earth ( Similar to the first movement, while raising the hands, one hand is directed upwards towards the sky and the other hand is directed towards the ground, turn the head and look back, shake the head and shake the tail (This movement regulates the functions of the heart and lungs, facilitates relaxation by relaxing the sympathetic nervous system, and helps emotional imbalances in the body). It is said that it removes the stagnation of Qi and eliminates the numbness and malaise in the legs. Its main purpose is to eliminate excessive heat in the heart), bending the waist down and holding the feet, punching, looking angry and shaking the ground by heeling will be done respectively.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study
* Having a complaint of urinary incontinence
* Being a woman between the ages of 45-55
* Being communicable
* Having a device (phone, tablet, computer) that can participate in online conversations
* Being in the premenopausal period

Exclusion Criteria:

* Women who do not complain of urinary incontinence
* Women in menopause
* Women who left unanswered questions on their scale forms

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Psychological Well-Being Scale | 4 month
  It was developed by Diener et al. to measure socio-psychological well-being as a complement to existing well-being measurements. The adaptation of the scale into Turkish was carried out by Telef. Factor loadings of the scale items were calculated between .54 and .76. The Cronbach's alpha internal consistency coefficient obtained in the reliability study of the scale was calculated as .80. All items are worded positively. Scores range from 8 to 56.
Incontinence Quality of Life Scale | 4 month
  It was developed by Wagner et al. in 1996 in America to determine the quality of life of patients with urinary incontinence. However, the scale was revised by Patrick et al. in 1999, and during the creation of the European versions, six questions were removed and the number of questions was reduced to 22 by evaluating the psychometric measurements. In our country, the validity and reliability of I-QOL was determined by Özerdoğan. It is converted to a scale value up to 100. Higher scores indicate a better level of quality of life than lower scores.

CONTACTS AND LOCATIONS:
Overall Officials: TUBA YILMAZ BULUT, Dr., Study Chair — Kocaeli University; Aynur ATAMAN KUFACI, Lecturer, Study Chair — Sinop University
Locations (1):
- Tuba Yilmaz Bulut, Kocaeli, Turkey (Türkiye)

REFERENCES:
- [Background] Wagner TH, Patrick DL, Bavendam TG, Martin ML, Buesching DP. Quality of life of persons with urinary incontinence: development of a new measure. Urology. 1996 Jan;47(1):67-71; discussion 71-2. doi: 10.1016/s0090-4295(99)80384-7. PMID 8560665
- [Background] Telef BB. Psychological Well-Being Scale (PIOO): Adaptation to Turkish, Validity and Reliability Study. Hacettepe Faculty of Education Journal, 2013; 28(3):374-384
- [Background] Diener E, Wirtz D, Tov W, Kim-Prieto C, Choi D, Oishi S, Biswas-Diener R. New well-being measures: Short scales to assess flourishing and positive and negative feelings. Social Indicators Research, 2010; 97: 143-156.
- [Background] Özerdoğan N, Kızılkaya NB. Prevalence, risk factors, and impact on quality of life of urinary incontinence in women aged 20 and over in Eskişehir, Bilecik, Afyon, Kütahya provinces. Journal of Nursing 2003; 13:37-50.